CLINICAL TRIAL: NCT07367919
Title: The Effect of a Digital Literacy Program on Problematic Internet Use, Emotion Regulation, and Loneliness in Adolescents: A Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Sümeyra Demireli, PhD student, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: B.30.2.ATA.0.01.00/399
Record Dates: First submitted 2025-12-10; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Healthy Adolescents
Keywords: Digital Literacy; Problematic Internet Use; Emotion Regulation; Loneliness
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Intervention Model Description: The study population consists of 9th, 10th, and 11th-grade students (N=2,578) attending secondary schools in Bayburt. Stratified sampling will be used to ensure homogeneity among classes, and experimental and control groups will be determined using a simple random method. Randomization will be conducted through random.org, and groups will be finalized before the eight-week training program. The study will be conducted at two different schools to prevent interaction between groups, and the control group will receive a two-week post-training program. Due to the nature of the study, blinding of the researcher will not be possible. Data will be collected by an independent interviewer, and statistical blinding will be applied. Sample size was calculated using G*Power 3.1.9.4 with α=0.05, power=0.85, and effect size=0.80. Approximately 32 students were planned for each group. The study is a randomized controlled trial with a pretest-posttest design.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be unaware of their group assignment. The intervention provider (researcher) will not be unaware of the nature of the educational intervention. Data collection will be conducted by an independent evaluator unaware of group assignment. Additionally, a data analyst will conduct statistical analysis unaware of group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Active Comparator): Participants in this group will participate in an eight-week positive youth development-based digital literacy program. The program includes in-person sessions with interactive exercises on digital literacy, problematic internet use, emotion regulation, and loneliness.
  Interventions: Other: DIGITAL LITERACY PROGRAM
- control group (No Intervention): Participants in this group will not receive any program during the study. Following the post-test measurements, they will receive two weeks of digital literacy training.

INTERVENTIONS:
Other: DIGITAL LITERACY PROGRAM — This intervention is an eight-week, face-to-face, Positive Youth Development-Based Digital Literacy Program designed specifically for adolescents. It includes interactive sessions, discussions, and exercises that address digital literacy, problematic internet use, emotion regulation, and loneliness. The program differs from other digital literacy interventions because it integrates positive youth development principles and focuses on both online behavior and emotional skills.
  Arms: experimental group

SUMMARY:
The purpose of this study is to examine the effects of a digital literacy program on problematic internet use, emotion regulation, and loneliness among adolescents. The study aims to answer the following key questions:

* Does a digital literacy program for adolescents affect problematic internet use, emotion regulation skills, and loneliness?
* What is the effect of a digital literacy program for adolescents on the level of problematic internet use?
* What is the effect of a digital literacy program for adolescents on emotion regulation skills?
* What is the effect of a digital literacy program for adolescents on loneliness? Researchers will conduct pretest and posttest evaluations in the experimental and control groups to determine the effects of the digital literacy program on problematic internet use, emotion regulation, and loneliness in adolescents. Participants in the experimental group who meet the inclusion criteria will receive 8 weeks of positive youth development-based digital literacy training, 40 minutes per week. After the posttest measurements are completed, the intervention group will receive 2 weeks of digital literacy training.

DETAILED DESCRIPTION:
Digital literacy is the process of developing individuals' access to accurate information, critical evaluation, ethical and responsible use, self-management, and social interaction skills. Digital media has become an indispensable part of life today. Individuals interact intensively with digital media, especially during adolescence, a period when interaction with the outside world intensifies, shapes an individual's identity, and heightens emotional awareness. During this critical developmental period, inadequate access to accurate information, critical thinking, and self-regulation skills pave the way for adolescents' problematic internet use. Problematic internet use negatively impacts individuals' academic success, friendships, and physical and mental health.

Emotion regulation, one of the most important skills for coping with risky situations that may arise from problematic internet use, supports adolescents' adaptability and is an effective skill in preventing negative digital interactions. Weak emotion regulation skills can make adolescents more vulnerable to negative digital interactions. Furthermore, increased time spent online and a decrease in face-to-face interactions can reinforce feelings of loneliness.

The program, developed with a positive youth development perspective, aims to increase adolescents' awareness of digital literacy, improve their emotion regulation skills, and reduce feelings of loneliness. The program is expected to provide important data for developing evidence-based intervention approaches for digital literacy within the scope of preventive mental health services in nursing, and particularly for nurses to assume more active roles in school-based preventive mental health services.

ELIGIBILITY:
Inclusion Criteria:

* Agreeing to participate in a face-to-face education program
* Obtaining written consent from students and parents
* Attending school during the study period
* Being a 9th, 10th, or 11th-grade student
* Scoring 52 or higher on the Generalized Problematic Internet Use Scale 2

Exclusion Criteria:

* Not completing the measurements and applications
* Not being able to participate in the program due to health or special circumstances
* Changing schools for any reason
* Being a 12th grade student
* Having previously received digital literacy training

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 64 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in Generalized Problematic Internet Use (GPIU-2) Scores | 8 weeks (baseline to post-intervention)
  The Turkish adaptation of the Generalized Problematic Internet Use Scale 2 (GPIUS2) will be used in the research. The scale consists of four subdimensions and 15 items, namely online social interaction preference, emotion regulation, inadequate self-regulation, and negative consequences. It is scored using a 5-point Likert-type scale with the values of "Strongly Disagree," "Disagree," "Undecided," "Agree," and "Strongly Agree." Caplan did not report a cutoff point for the original Generalized Problematic Internet Use Scale 2. In the study conducted by Machimbarrena et al., an ROC curve analysis was performed to determine the cutoff point for GPIUS2, and a score of 52 was recommended to distinguish problematic and non-problematic internet users.
Change in Emotion Regulation Scores | 8 weeks (baseline to post-intervention)
  The Emotion Regulation Scale for Adolescents is a tool for assessing adolescents' emotion regulation with four subdimensions: internal functional emotion regulation, internal dysfunctional emotion regulation, external functional emotion regulation, and external dysfunctional emotion regulation. The scale consists of a total of 18 items and is scored using a 5-point Likert-type scale: "Never (1), Rarely (2), Sometimes (3), Most of the time (4), and Always (5). Item response scores for each subdimension are calculated individually and indicate the individual's frequency of using the relevant emotion regulation method. The subdimension with the highest total score is the individual's most frequently used emotion regulation method. There are no reverse-scored items.
Change in Adolescent Loneliness Scores | 8 weeks (baseline to post-intervention)
  The single-dimensional scale, applied to adolescents aged 14-19, consists of 7 items and is scored with a 4-point Likert-type scale of "(1) Never, (2) Rarely, (3) Sometimes, and (4) Always." Item 5 of the scale is reverse-scored. The highest score that can be obtained from the scale is 28, while the lowest is 7. Higher scores indicate higher feelings of loneliness. The Cronbach's alpha internal consistency coefficient of the scale was found to be α=0.74. The test-retest reliability of the UYÖ-SF, administered to 64 high school students at a two-week interval, was found to be r=0.84.

CONTACTS AND LOCATIONS:
Overall Officials: Sümeyra DEMİRELİ, PhD student, Principal Investigator — Ataturk University; Hatice DURMAZ, Associate Professor, Study Director — Ataturk University
Locations (1):
- Bayburt Milli İrade Anadolu Lisesi, Bayburt Fen Lisesi, Bayburt, Bayburt, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared, as the participant consent form states that the data will be used only for this study.